CLINICAL TRIAL: NCT06670326
Title: Imagery Rescripting As a Treatment for Pathological Affective Dependence: Helping Victims Break Free from Abusive Relationships
Brief Title: Imagery Rescripting for Pathological Affective Dependence and Intimate Partner Violence
Acronym: ImRs-PAD
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Amsterdam (Other)
Collaborators: VU University of Amsterdam (Other); Stichting Achmea Slachtoffer en Samenleving (Other)
Responsible Party: Principal Investigator, Erica Pugliese, Principal Investigator, University of Amsterdam
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: FMG-10908
Record Dates: First submitted 2024-10-17; First posted 2024-11-01 (Actual); Last update posted 2024-11-01 (Actual); Status verified 2024-10

CONDITIONS: Pathological Affective Dependence
Keywords: Imagery Rescripting; Pathological Affective Dependence; Treatment; intimate partner violence

STUDY DESIGN:
Intervention Model Description: Multiple baseline case series design: by randomizing participants to different lengths of waitlist (baseline) and comparing means and slopes of weekly reported Pathological Affective Dependence severity and mental health measures, the effectiveness of the treatment is tested.
Masking Description: The investigator will not have access to assignment of participants to waitlist length and the data until data collection is complete.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Baseline-Preparation-Imagery Rescripting-Post Treatment (Experimental): Each participant follows this sequence: (1) 5-9 weeks waitlist during which no treatment is offered; (2) 4 weekly preparatory sessions. During these sessions the rationale of ImRs will be explained in more detail and a list of painful (childhood) memories to be addressed with ImRs is to be compiled, based on any further input from the patient; and a case conceptualization is made; (3) 12 sessions (45-60 minutes) of ImRs will be offered to participating patients. The ImRs treatment will be based upon the protocol described by Arntz & Weertman (1999). This protocol can be modified to tailor the needs of this study more specifically. (4) After end of active treatment (ImRs) 4 weeks follow during which only weekly assessments are done.
  Interventions: Behavioral: Imagery Rescripting

INTERVENTIONS:
Behavioral: Imagery Rescripting — Experimental: Baseline-Preparation-Imagery Rescripting-Post Treatment Each participant follows this sequence: (1) 5-9 weeks waitlist during which no treatment is offered; (2) 4 weekly preparatory sessions. During these sessions the rationale of ImRs will be explained in more detail and a list of painful (childhood) memories to be addressed with ImRs is to be compiled, based on any further input from the patient; and a case conceptualization is made; (3) 12 sessions (45-60 minutes) of ImRs will be offered to participating patients. The treatment for PAD will be based upon the protocol described by Arntz & Weertman (1999); (4) After end of active treatment (ImRs) 4 weeks follow during which only weekly assessments are done.
  Other Names: ImRs

SUMMARY:
The goal of this multiple baseline case series study is to evaluate the effectiveness of Imagery Rescripting for Pathological Affective Dependence (PAD) in victims of Intimate Partner Violence (IPV). The primary research questions are:

Does Imagery Rescripting reduce PAD and/or commitment to the abusive relationship after separation? Does Imagery Rescripting also reduce traumatic symptoms? Does Imagery Rescripting improve general mental health, self-compassion, and resilience in IPV victims? Participants will undergo a waiting period of 5-9 weeks (to assess time effects without treatment), followed by 4 weekly preparation sessions, 12 weekly Imagery Rescripting sessions, and 1 month of post-treatment.

Throughout the study, participants will rate the severity of PAD and relational commitment on a weekly basis. They will also complete more detailed questionnaires assessing mental health, traumatic symptoms, resilience, and self-compassion before each phase, at 1 month post-treatment, 3 months post-treatment, and during follow-ups at 6 and 12 months.

DETAILED DESCRIPTION:
In this multiple baseline case series study, the effectiveness of Imagery Rescripting (ImRs) as a treatment for Pathological Affective Dependence (PAD) in victims of Intimate Partner Violence (IPV) will be evaluated. Eighteen victims of IPV with PAD will be randomized to different waitlist lengths (5-9 weeks), after which they will enter a 4-session preparation phase (4 weeks), followed by 12 weekly sessions of ImRs. Follow-up assessments will take place at 4 weeks, 6 months, and 12 months post-treatment.

The primary outcomes are:

PAD severity, which will be assessed weekly using the Pathological Affective Dependence Scale.

Relational commitment, measured using a validated scale. The hypothesis is that primary outcomes will show greater reductions during the treatment phase compared to the waitlist or preparation phases and will either stabilize or show further improvement post-treatment.

Similarly, secondary outcomes such as general mental health (measured by the Patient Health Questionnaire, PHQ-9), resilience (assessed with the The Brief Resilience Scale (RSb), and self-compassion (assessed with the Self-compassion Scale short (SCs) are expected to show the most significant improvements from pre- to post-treatment, with minimal changes during baseline, preparation, and post-treatment phases.

The results will be analyzed using multilevel analysis, pooling the effects across individual cases. In addition, participants will be interviewed 4 weeks post-treatment to gather qualitative feedback on their experiences with the treatment.

ELIGIBILITY:
Inclusion Criteria:

* Experience of IPV (from a clinical interview)
* Pathological Affective Dependence scale (PADS - Trait, State). As a prerequisite for PAD treatment and study participation, victims of IPV are required to establish a contact with the anti-violence center or shelters to receive co-assistance. The anti-violence center will take care of his/her physical safety and legal aspects.

Exclusion Criteria:

* Comorbidity with the following diagnoses: psychosis, schizophrenia, bipolar disorder (conditions derived from a clinical interview or previous diagnostic reports), dissociative disorders (Dissociative Experience Scale, DES).
* Organic brain disease
* Intelligence Quotient (IQ) < 80
* High risk of self-harm or suicide
* Current substance abuse severe level
* Start of new medication within 2 months before beginning the study (medication used for longer periods can be continued; patients are requested to keep medication stable during the course of the study)
* Having received ImRs (either as a stand-alone or embedded in a greater treatment such as cognitive behavior therapy (CBT) or schema therapy) within the last year
* No other evidence-based treatment of MDD is allowed during the study.
* Not able to plan enough time for weekly therapy sessions (45-60 minutes); weekly measurements (estimate of 5 minutes) and other measurements (estimate of 20 minutes); and the qualitative post-treatment interview (estimate of 60 minutes) during the study period.

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Estimated)
Dates: Start 2025-02-01 (Estimated); Primary Completion 2025-05 (Estimated); Study Completion 2026-02 (Estimated)

PRIMARY OUTCOMES:
Pathological Affective Dependence Scale (PADS) | 22-32 weeks plus 3, 6 and 12 months follow-ups
  The PADS (Pugliese et al., 2024) is a 17-item Likert-type scale designed to assess both the state and trait manifestations of Pathological Affective Dependence (PAD), particularly focusing on the factors that compel individuals to remain in abusive relationships. These factors include internal conflict, the inability to separate from an abusive partner, and experiences of partner abuse. The scale is administered twice, with instructions tailored to measure both state and trait PAD. Each item is rated on a 5-point Likert scale, where 1 = not at all, 2 = slightly, 3 = sometimes, 4 = often, and 5 = always.
Relational Commitment (RC) | 22-32 weeks plus 3, 6 and 12 months follow-ups
  The seven items of the Relationship Commitment scale (Rusbult, Martz, & Agnew, 1998) include the following items: for example, "I am committed to maintaining my relationship with my partner"; "I want our relationship to last for a very long time"; "I feel very attached to our relationship". Responses are rated on an 8-point scale ranging from 1 (Do not agree at all) to 8 (Agree completely).

SECONDARY OUTCOMES:
Patient Health Questionnaire (PHQ-9 and PHQ-15) | before baseline, before preparatory sessions, before ImRs treatment, 4 weeks after ImRs treatment, 3, 6 and 12 months follow-ups
  Patient Health Questionnaire-15 (PHQ-15) is a 15-item self-report tool to measure somatic symptoms. Items responses ranged from 0 (not at all) to 2 (bothered a lot). The total score is calculated by adding all item responses, and scores of 5, 10, and 15 represent cutpoints for low, medium, and high somatic symptom severity, respectively (Spitzer et al., 1999).
  - Patient Health Questionnaire-9 (PHQ-9) is a 9-item self-report tool to measure depression symptoms. Item responses ranged from 0 (not at all) to 3 (nearly every day). The total score is calculated by adding all item responses, and scores of 5, 10, 15, and 20 represent cutpoints for mild, moderate, moderately severe, and severe depression, respectively (Kroenke et al., 2001)
Self-compassion Scale short (SCs) | before baseline, before preparatory sessions, before ImRs treatment, 4 weeks after ImRs treatment, 3, 6 and 12 months follow-ups
  Self-Compassion Scale-Short Form (SCS-SF) is a 12-item tool to measure self-compassion. It is composed of six dimensions, each with two items: Self-Kindness (SK), Self-Judgment (SJ), Common Humanity (CH), Isolation (I), Mindfulness (M), and Over-Identification (OI). Items responses ranged from 1 (almost never) to 5 (almost always). Subscale scores are computed by adding item scores, and a total self-compassion score is calculated by reversing the negative subscale items and then adding all subscale scores. Higher scores correspond to higher self-compassion. The internal consistencies ranged between 0.54 to 0.75, and the total Cronbach's alpha was 0.87 (Raes et al., 2011).
Psychological General Well-Being Index (PGWB-S) | before baseline, before preparatory sessions, before ImRs treatment, 4 weeks after ImRs treatment, 3, 6 and 12 months follow-ups
  Patient Health Questionnaire-15 (PHQ-15) is a 15-item self-report tool to measure somatic symptoms. Items responses ranged from 0 (not at all) to 2 (bothered a lot). The total score is calculated by adding all item responses, and scores of 5, 10, and 15 represent cutpoints for low, medium, and high somatic symptom severity, respectively (Spitzer et al., 1999).
  - Patient Health Questionnaire-9 (PHQ-9) is a 9-item self-report tool to measure depression symptoms. Item responses ranged from 0 (not at all) to 3 (nearly every day). The total score is calculated by adding all item responses, and scores of 5, 10, 15, and 20 represent cutpoints for mild, moderate, moderately severe, and severe depression, respectively (Kroenke et al., 2001)
The Brief Resilience Scale (RSb) | before baseline, before preparatory sessions, before ImRs treatment, 4 weeks after ImRs treatment, 3, 6 and 12 months follow-ups
  Brief Resilience Scale (BRS): is a 6-item unidimensional tool to measure individual resilience levels. Three items are positively worded, and three are negatively worded. The total score was calculated by reversing items 2, 4, and 6 and then adding all items. Items responses ranged from 1 (strongly disagree) to 5 (strongly agree). Higher scores correspond to higher resilience. Internal consistency ranges from 0.80 to 0.91 (Smith et al., 2008).
Generalized Anxiety Disorder 7-item Scale (GAD-7) | before baseline, before preparatory sessions, before ImRs treatment, 4 weeks after ImRs treatment, 3, 6 and 12 months follow-ups
  Generalized Anxiety Disorder 7-item Scale (GAD-7) is a 7-item self-report tool to measure anxiety symptoms. Item responses ranged from 0 (not at all) to 3 (nearly every day). The total score is calculated by adding all item responses, and scores of 5, 10, and 15 represent cutpoints for mild, moderate, and severe anxiety, respectively (Spitzer et al., 2006)

OTHER OUTCOMES:
patients' experiences | 4 weeks after end of treatment
  with a semi-structured interview, participants will be interviewed 4 weeks after treatment. A qualitative analysis will be used.

CONTACTS AND LOCATIONS:
Overall Officials: Erica Pugliese, PhD, Principal Investigator — University of Amsterdam
Locations (3):
- Associazione Italiana Di Psicoterapia Cognitiva - Aipc, Bari, Italy, Italy
- Netherlands (2):
  - Sterk Huis, Amsterdam, Goirle
  - University of Amsterdam, Amsterdam

IPD SHARING:
Plan to Share IPD: No
because of privacy regulations individual patient data cannot be shared, unless the European Union (EU) regulations on data protection are guaranteed.